CLINICAL TRIAL: NCT02531542
Title: Evaluation of Rapid Emergency Echography for Acute Dyspnoea for the Diagnosis of Acute Left-sided Heart Failure in Elderly Subjects Admitted to the Emergency Room (READ Protocol)
Brief Title: Evaluation of Rapid Emergency Echography for Acute Dyspnoea
Acronym: READ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Centre Hospitalier Germon et Gauthier (Unknown); University Hospital, Clermont-Ferrand (Other); Centre Hospitalier de PAU (Other); University Hospital, Strasbourg, France (Other); Centre Hospitalier Général de Toulon (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: N/2014/69
Record Dates: First submitted 2015-08-12; First posted 2015-08-24 (Estimated); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Acute Dyspnea

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- READ echography (Other)
  Interventions: Device: Echocardiography according to the READ method.

INTERVENTIONS:
Device: Echocardiography according to the READ method. — * Echocardiography will be performed before any therapy is initiated by a fully trained operator, according to the READ method. The results of this ultrasound will not be communicated to the clinician managing the patient in the emergency room.
  * A blood sample will be taken during the routine work-up for centralized evaluation of NT-proBNP levels.

SUMMARY:
Elderly people constitute the largest proportion of emergency room patients, representing 12% of all emergency room admissions. The need for diagnostic tests or therapeutic interventions is much greater in this patient population. Cardiovascular diseases and symptoms represent 12% of the causes for emergency room admission, and patients suffering from cardiovascular disease are those whose emergency room visit lasts longest.

The diagnostic approach in the emergency room in elderly patients admitted for acute dypsnoea is complex, and early identification of acute left-sided heart failure (ALSHF) is vital as it has an impact on prognosis. The clinical signs are difficult to interpret, and are non-specific, particularly at the acute phase and in elderly or obese patients. Indeed, some authors have reported up to 50% of diagnostic errors in elderly patients.

Measure of the blood concentration of a natriuretic peptide allows a quick diagnosis. However, peptides suffer from several limitations, particularly in situations that are often encountered in elderly patients, such as sepsis, renal failure, acute coronary syndrome, pulmonary embolism, chronic respiratory failure, atrial fibrillation and high body mass index. Diagnostic performance deteriorates with increasing age, and there is a significant increase in this grey-zone in patients aged ≥75 years. In critical situations in elderly patients, assessment of natriuretic peptides serve mainly to rule out a diagnosis of left heart failure.

Some authors have suggested using lung ultrasound in the initial work-up of acute respiratory failure, since some specific profiles are known to be related to the presence of interstitial oedema, reflecting impaired left heart function (e.g. presence of B lines). These studies were performed in the context of intensive or critical care, but data are sparse regarding the application of this approach in the emergency room.

The hypothesis is that the diagnostic accuracy of a targeted and quick echographic approach, namely the READ method (Rapid Echography for Acute Dyspnoea), comprising targeted lung ultrasound combined with isolated measure of transmitral flow, would be superior to that of NT-proBNP assessment for the diagnosis of ALSHF in elderly patients (≥75 years) admitted to the emergency department.

DETAILED DESCRIPTION:
The number of emergency room visits is constantly increasing, and it is therefore necessary to minimize the duration of each visit, thereby increasing the efficacy of the diagnostic process, leading to quicker orientation of each patient for appropriate care. In this context, accurate triage and a quick initial diagnostic work-up are of paramount importance in achieving this goal.

Elderly people constitute the largest proportion of emergency room patients, representing 12% of all emergency room admissions. The need for diagnostic tests or therapeutic interventions is much greater in this patient population, with 4 out of 5 patients requiring such measures. Indeed, elderly persons often suffer from multiple diseases that require a greater number of tests (source: Direction de la recherche, des études, de l'évaluation et des statistiques (DREES), emergency room survey) (1).

Cardiovascular diseases and symptoms represent 12% of the causes for emergency room admission, and patients suffering from cardiovascular disease are those whose emergency room visit lasts longest. Indeed, almost 50% of patients with cardiovascular disease stay more than 4 hours in the emergency room, according to a French national survey published in July 2014.

The diagnostic approach in the emergency room in elderly patients admitted for acute dypsnoea is complex, and early identification of acute left-sided heart failure (ALSHF) is vital as it has an impact on prognosis.

Acute dyspnoea and acute respiratory insufficiency are frequent causes of admission to the emergency room. The etiological diagnosis is difficult, especially in elderly patients who often have a history of cardio-respiratory disease (2)(3)(4)(5). In this specific population, there are often numerous comorbidities, such as chronic respiratory failure, chronic renal failure, and ischemic heart disease (6). In addition, acute respiratory insufficiency can be caused by a range of distinct pathologies, such as acute heart failure, pneumonia, exacerbation of chronic obstructive pulmonary disease (COPD), pleural effusion or pulmonary embolism. There is thus clearly a pressing need for an accurate and early diagnosis of the correct etiology in these patients, particularly to identify ALSHF, a condition that requires immediate initiation of appropriate therapy in order to improve prognosis. In these patients, studies have shown that inappropriate or delayed therapy in the emergency room is an independent predictor of death (2)(3)(7).

The European Society of Cardiology (ESC) recently published a review of the standard diagnostic methods for ALSHF, describing the advantages and limitations of each (clinical examination, electrocardiogram (ECG), chest x-ray, NT-proBNP assessment) (8).

The clinical signs are difficult to interpret, and are non-specific, particularly at the acute phase and in elderly or obese patients (9). Indeed, some authors have reported up to 50% of diagnostic errors in elderly patients (10).

Chest x-ray, which is usually performed in the emergency room, is not specific because of the conditions in which it is performed in emergency situations. Generally, the pre-requisites for proper implementation are not fully respected because of the emergency nature of the exam, and chest x-ray is therefore primarily useful for differential diagnosis only (8).

Early echocardiography is recommended in patients presenting to the hospital in an emergency with suspected heart failure (HF) and acute onset of symptoms. Imaging techniques play a central role in the diagnosis of HF and in guiding treatment. Among the several imaging modalities available, echocardiography is the method of choice in patients with suspected HF for reasons of accuracy, availability (including portability), safety and cost. The term echocardiography is used here to refer to all cardiac ultrasound imaging techniques, including two- or three-dimensional echocardiography, pulsed and continuous wave Doppler, colour flow Doppler, and tissue Doppler imaging. For assessment of left ventricular systolic and diastolic dysfunction, no single echocardiographic parameter is sufficiently accurate and reproducible to be used in isolation. Therefore, a comprehensive echocardiographic examination incorporating all relevant two-dimensional and Doppler data is recommended. This should include the evaluation of both structural and functional abnormalities.

However, this type of specialised echocardiography is not routinely available in most emergency rooms. In routine practice, systematic specialised echocardiography by a cardiologist for all cases of acute respiratory failure is not feasible due to the lack of trained operators. Indeed, training in specialised echocardiography is not a pre-requisite to become a qualified emergency room physician in France. Lastly, specialised echocardiography exams are time-consuming and incompatible with the need to manage the vast flow of patients through a busy emergency room.

An alternative approach to diagnosis is to measure the blood concentration of a natriuretic peptide, a family of hormones secreted in increased amounts when the heart is diseased or the load on any chamber is increased (11)(12)(13)(14)(15)(16). However, peptides suffer from several limitations, particularly in situations that are often encountered in elderly patients, such as sepsis, renal failure, acute coronary syndrome, pulmonary embolism, chronic respiratory failure, atrial fibrillation and high body mass index (17). Diagnostic performance deteriorates with increasing age, and there is a significant increase in this grey-zone in patients aged ≥75 years (8)(16)(18)(19). In critical situations in elderly patients, assessment of natriuretic peptides serve mainly to rule out a diagnosis of left heart failure (8)(16)(19).

Some authors have suggested using lung ultrasound in the initial work-up of acute respiratory failure (20)(21)(22)(23)(24)(25)(26), since some specific profiles are known to be related to the presence of interstitial oedema, reflecting impaired left heart function (e.g. presence of B lines) (27)(28). These studies were performed in the context of intensive or critical care, but data are sparse regarding the application of this approach in the emergency room.

In a preliminary, single-centre study, the utility of a quick transthoracic echography approach was investigated, namely the READ method (Rapid Echography for Acute Dyspnoea), which associated targeted lung ultrasound and measure of transmitral flow in 51 patients aged ≥75 years. When performed at the patient's admission to the emergency room, the READ method was showed to have a sensitivity of 95% for the identification of ALSHF. Indeed, analysis of transmitral flow is easily available by transthoracic echography. The presence of a "restrictive" pattern in case of acute dypsnoea is associated with the existence of ALSHF (29)(30)(31)(32)(33).

Echography is a diagnostic tool whose use in the emergency room is increasing exponentially. For example, the "Focused Assessment with Sonography in Trauma" (FAST) ultrasound assessment technique in trauma patients has become the cornerstone of initial triage in trauma patients. The idea is to use targeted ultrasound, not necessarily performed by a specialist, to achieve accurate triage of patients in only a few minutes to guide subsequent diagnostic and therapeutic approaches.

There is a paucity of well-conducted studies in the literature evaluating the utility of targeted chest ultrasound in the diagnostic work-up of acute dyspnoea in elderly patients admitted to the emergency department. There currently exists no consensus regarding the use of echography in these patients, and its use largely depends on the competency and availability of operators in the emergency, in the absence of formal evidence proving its utility. Biomarkers such as brain natriuretic peptide (BNP) or NT-proBNP lack sensitivity in this age-category of patients, although they are widely used in routine practice given the impossibility of rapid, and 24/7 access to specialised echocardiography.

In this context, the study hypothesis is that the diagnostic accuracy of a targeted and quick echographic approach, namely the READ method (Rapid Echography for Acute Dyspnoea), comprising targeted lung ultrasound combined with isolated measure of transmitral flow, would be superior to that of NT-proBNP assessment for the diagnosis of ALSHF in elderly patients (≥75 years) admitted to the emergency department.

ELIGIBILITY:
Inclusion Criteria:

Admission to the Emergency Department Age ≥ 75 years

AND criteria of acute dyspnoea:

* Breathe rate ≥ 25 cycles/minute
* or PaO2 ≤ 70 mmHg
* or SpO2 ≤ 92% in room air
* or PacO2 ≥ 45 mmHg and pH ≤ 7.35 AND Electrocardiogram in sinus rhythm or in atrial fibrillation at admission

Exclusion Criteria:

* Shock i.e. : systolic arterial pressure <90mmHg; or reduction >40mmHg or >30% of usual arterial pressure; or Mean Arterial Pressure <65mmHG.
* Acute respiratory distress ie : Respiratory rate >30cpm, use of accessory respiratory muscles, SpO2 <90% when O2 therapy is required, impaired consciousness,
* Presence of acute coronary syndrome on the ECG
* Other obvious etiological diagnosis (pneumothorax, clinical and radiological manifestations of pneumonia)
* Cardiological or respiratory medicine therapies initiated before the READ approach could be put in place (at patient's home, pre-hospital and/or in the emergency department) i.e.. diuretic, vasoactive drugs (nitrovasodilator, sympathomimetic and cardiotonic drugs, vasodilators and vasoconstrictors); or Continuous Positive Airway Pressure (CPAP); or invasive or non-invasive ventilation.
* Patient not affiliated to or beneficiary of the French social security system
* Protected people (pregnant and lactating women, guardianship, curatorship, under the protection of justice)Subjects in the exclusion period after participation in another clinical trial, or as listed in the national database of health research volunteers

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 461 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
To demonstrate the superiority of the READ method over assessment of NT-proBNP for the diagnosis of acute left-sided heart failure in patients aged ≥75 years admitted to the emergency department for acute dyspnoea. | 1 day
  The diagnosis of ALSHF will be established post hoc by two experts based on a specialised echocardiography performed within 7 days after inclusion, or before discharge (whichever occurs first) and on the patient's medical file.
  The presence of ALSHF using the READ method is defined as presence of diffuse B-lines on lung ultrasound, combined with a restrictive pattern on analysis of transmitral profile.
  A diagnosis of ALSHF will be retained if the NT-proBNP level is greater than the threshold value of 1800 pg/mL, which is the appropriate threshold for patients aged >75 years.

SECONDARY OUTCOMES:
To evaluate the utility of the combination of the READ method and assessment of NT-proBNP for the diagnosis of ALSHF. | 1 day
  The diagnostic value of the test, assessed in terms of sensitivity and specificity, will be calculated based on the optimal combination of the results of the two tests, namely the READ method and NT-proBNP assessment.
To assess the potential influence of patients characteristics (age, sex, clinical presentation) on the diagnostic performance of each method of diagnosis (READ and NT-proBNP assessment). | 1 day
  We will investigate the possible presence of a spectrum effect, mainly in terms of age and gender, in the population.
To evaluate agreement between the results of the READ approach interpreted immediately in the emergency setting, vs deferred evaluation (outside the emergency setting) of the same images by a different operator. | 1 day
  We will evaluate agreement between the results of the READ approach interpreted immediately in the emergency setting, vs deferred evaluation (outside the emergency setting) of the same images by a different expert operator.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - University Hospital of Clermont-Ferrand, Clermont-Ferrand, Auvergne
  - University Hospital of Strasbourg, Strasbourg, Grand Est
  - Centre hospitalier de Pau, Pau, Nouvelle-Aquitaine
  - University Hospital of Toulouse, Toulouse, Occitanie
  - Centre Hospitalier de Toulon, Toulon, Provence-Alpes-Côte d'Azur Region